CLINICAL TRIAL: NCT04950920
Title: Phase III Clinical Trial of Y-2 Sublingual Tablet in the Treatment of Acute Ischemic Stroke - a Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Clinical Trial
Brief Title: Phase III Clinical Trial of Y-2 Sublingual Tablets in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2020185
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-2 sublingual test group (Experimental): Y-2 sublingual tablets: Edaravone 30mg and d-borneol 6mg.
  Interventions: Drug: Y-2 sublingual tablets
- placebo group (Sham Comparator): 60 μg d-borneol
  Interventions: Drug: d-borneol

INTERVENTIONS:
Drug: Y-2 sublingual tablets — 30mg Edaravone+6mg d-borneo OR， Bid
  Arms: Y-2 sublingual test group
Drug: d-borneol — 60 μg d-borneol OR， Bid
  Arms: placebo group

SUMMARY:
At present, the treatment of acute ischemic stroke includes intravenous thrombolysis, intravascular interventional therapy (including arterial thrombolysis, mechanical thrombectomy, angioplasty and stent implantation), antiplatelet therapy, anticoagulant therapy, defibrasion therapy, volume expansion therapy, and neuroprotective therapy. Y-2 sublingual tablet is an innovative drug developed by Yantai yinuoyi Biomedical Technology Co., Ltd. with independent intellectual property rights. This product is a free radical scavenger and inflammatory protein expression inhibitor. It can clear hydroxyl free radical (COH), nitric oxide free radical (no) and peroxynitrite ion (onoa), and inhibit the expression of tumor necrosis factor-A (TNF-a), interleukin IP (IL-1 (3), cyclooxygenase-2 (COX-2) and inducible nitric oxide synthase (iNOS) and other inflammatory related proteins induced by cerebral ischemia. By clearing the excessive free radicals produced in the brain tissue during ischemia and reperfusion and inhibiting the secondary inflammatory reaction, we can reduce the damage of free radicals and inflammatory reaction to the brain tissue, block the pathological change process caused by cerebral ischemia from two ways, and play a synergistic therapeutic role in cerebral ischemia injury.

DETAILED DESCRIPTION:
At present, the treatment of acute ischemic stroke includes intravenous thrombolysis, intravascular interventional therapy (including arterial thrombolysis, mechanical thrombectomy, angioplasty and stent implantation), antiplatelet therapy, anticoagulant therapy, defibrasion therapy, volume expansion therapy, and neuroprotective therapy. Y-2 sublingual tablet is an innovative drug developed by Yantai Yinuoyi Biomedical Technology Co., Ltd. with independent intellectual property rights. This product is a free radical scavenger and inflammatory protein expression inhibitor. It can clear hydroxyl free radical (COH), nitric oxide free radical (no) and peroxynitrite ion (onoa), and inhibit the expression of tumor necrosis factor-A (TNF-a), interleukin IP (IL-1 (3), cyclooxygenase-2 (COX-2) and inducible nitric oxide synthase (iNOS) and other inflammatory related proteins induced by cerebral ischemia. By clearing the excessive free radicals produced in the brain tissue during ischemia and reperfusion and inhibiting the secondary inflammatory reaction, we can reduce the damage of free radicals and inflammatory reaction to the brain tissue, block the pathological change process caused by cerebral ischemia from two ways, and play a synergistic therapeutic role in cerebral ischemia injury.

ELIGIBILITY:
Inclusion Criteria:

-

Those who meet all of the following requirements:

1. Age ≥ 18 years old and ≤ 80 years old, regardless of gender;
2. After the onset of the disease, the National Institutes of Stroke Scale score: 6 ≤ NIHSS ≤ 20, and the sum of the fifth upper limb score and the sixth lower limb score was ≥2;
3. The onset time is within 48 hours (including 48 hours);
4. Patients diagnosed as ischemic stroke according to "key points for diagnosis of all kinds of major cerebrovascular diseases in China 2019", with good prognosis after the first attack or the last attack (MRS score ≤ 1 before this attack);
5. The informed consent approved by the ethics committee was voluntarily signed by the patient or his legal representative.

Exclusion Criteria:

-

Those who meet any of the following items:

1. Intracranial hemorrhagic diseases seen in head imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc; If it is only oozing blood, the researcher can judge whether it is suitable for inclusion;
2. Severe disturbance of consciousness: the item score of La consciousness level of NIHSS was more than 1;
3. Transient ischemic attack (TIA);
4. Systolic blood pressure was still higher than 220mmhg or diastolic blood pressure was higher than 120mmhg after blood pressure control;
5. Patients with severe mental disorders and dementia;
6. Severe active liver diseases have been diagnosed, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc; Or ALT or AST > 2.0 × ULN;
7. Severe active kidney disease and renal insufficiency have been diagnosed; Or serum creatinine > 1.5 × ULN;
8. After the onset of the disease, the drugs with neuroprotective effect in the manual have been used;
9. Embolectomy or interventional therapy has been used or planned after the onset of the disease;
10. Complicated with malignant tumor or undergoing anti-tumor treatment; For the subjects diagnosed with malignant tumor after enrollment, whether to continue to participate in the study can be judged by the researcher and the willingness of the subjects;
11. Suffering from severe systemic diseases, the estimated survival time is less than 90 days;
12. Allergic to d-borneol or edaravone or excipients;
13. Patients during pregnancy, lactation and planned pregnancy;
14. Major operation history within 4 weeks before enrollment;
15. Have participated in other clinical studies or are participating in other clinical studies within 30 days before randomization;
16. The researcher thinks that it is not suitable to participate in this clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
mRS score ≤ 1 | 90 days after treatment initiation
  Whether patients with mRS(Modified Rankin Scale) score ≤ 1. Used to calculate the proportion of patients with mRS score ≤ 1.

SECONDARY OUTCOMES:
patients' mRS score | 90 days after treatment initiation
  patients' modified Rankin score
Good functional outcome | 90 days after treatment initiation
  Whether patients with mRS score ≤ 2. Used to calculate the proportion of good functional outcome (mRS ≤2)
change of NIHSS score | 14 after treatment initiation
  Change of NIHSS (National Institute of Health stroke scale) score from baseline to day 14 after randomization
NIHSS score≤1 on 14 day | 14 after treatment initiation
  Whether NIHSS (National Institute of Health stroke scale) score≤1 on 14 day. Used to calculate the proportion of NIHSS score≤1 on 14 day.
NIHSS score≤1 on 30 day | 30 after treatment initiation
  Whether NIHSS (National Institute of Health stroke scale) score≤1 on 30 day. Used to calculate the proportion of NIHSS score≤1 on 30 day.
NIHSS score≤1 on 90 day | 90 after treatment initiation
  Whether NIHSS (National Institute of Health stroke scale) score≤1 on 90 day. Used to calculate the proportion of NIHSS score≤1 on 90 day.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu Y, Wang A, Tang R, Li S, Tian X, Xia X, Ren J, Yang S, Chen R, Zhu S, Feng X, Yao J, Wei Y, Dong X, Ling Y, Yi F, Deng Q, Guo C, Sui Y, Han S, Wen G, Li C, Dong A, Sun X, Wang Z, Shi X, Liu B, Fan D. Sublingual Edaravone Dexborneol for the Treatment of Acute Ischemic Stroke: The TASTE-SL Randomized Clinical Trial. JAMA Neurol. 2024 Feb 19;81(4):319-26. doi: 10.1001/jamaneurol.2023.5716. Online ahead of print. PMID 38372981
- [Derived] Fu Y, Tang R, Chen R, Wang A, Ren J, Zhu S, Feng X, Fan D. Efficacy and safety of Y-2 sublingual tablet for patients with acute ischaemic stroke: protocol of a phase III randomised double-blind placebo-controlled multicentre trial. Stroke Vasc Neurol. 2024 Feb 27;9(1):90-95. doi: 10.1136/svn-2022-002014. PMID 37308251